CLINICAL TRIAL: NCT02553759
Title: Influence of the Actions Observed on Cervical Motion in Patients With Chronic Neck Pain. Randomized Controlled Trial
Brief Title: Observed Actions in Chronic Neck Pain
Acronym: ObACNPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AG Clinic (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Alfonso Gil Martínez, Physiothreapist. Master in Science, AG Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ObActions
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Pain
Keywords: observed action; range of motion; mirror neuron
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Effective movement (Experimental): This group will see a 1-minute video showing an individual performing a cervical rotation movement to each side, first 10 times towards the right and then 10 times towards the left. The movement will be performed effectively over the entire course of the cervical path, approximately 80º
  Interventions: Other: Actions observed
- Ineffective movement (Active Comparator): This group will see a 1-minute video showing an individual performing a cervical rotation movement ineffectively, without achieving the maximum cervical travel, performing approximately 40º. First, 10 movements towards the right will be performed and then 10 towards the left
  Interventions: Other: Actions observed

INTERVENTIONS:
Other: Actions observed — Patients observed movements without realize them. After this actions, movements will be imagined by patients

SUMMARY:
The aim of the present protocol is to prove if the observed actions (AOb) will improve the cervical range of motion (CROM) in patients with non-specific chronic neck pain (CNP). This study is a parallel-group double blind randomized clinical. Outcome measures were CROM, and pressure pain detection thresholds (PPDT) with a digital algometer. The follow-up will consist of three evaluations: pre- treatment, post-treatment and 10 minutes after second measurement (motor imagery).

ELIGIBILITY:
Inclusion Criteria:

* Non specific chronic neck pain
* Diagnosed by medical specialist

Exclusion Criteria:

* cervical osteoarthritis or polyarthrosis
* rheumatic disease
* history of cervical hernia
* whiplash syndrome
* surgery on the neck, face or shoulders,
* systemic disease, medical history of cancer
* significant trauma that the patient relates to their pain and/or refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Range of motion degrees | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Gil-Martínez, Master, Study Director — Hospital Universitario La Paz